CLINICAL TRIAL: NCT04464473
Title: cTBS/fMRI Study of Hierarchical Control in the PFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Derek Nee, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00000532; R01MH121509 (NIH)
Record Dates: First submitted 2020-06-12; First posted 2020-07-09 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Transcranial Magnetic Stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- FPl-TMS (Experimental): Transcranial magnetic stimulation to the lateral frontal pole. 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold.
  Interventions: Device: transcranial magnetic stimulation
- MFG-TMS (Experimental): Transcranial magnetic stimulation to the middle frontal gyrus. 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold..
  Interventions: Device: transcranial magnetic stimulation
- S1-TMS (Active Comparator): Transcranial magnetic stimulation to primary somatosensory cortex. 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold..
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.

SUMMARY:
The objective of this study is to examine the effect of transcranial magnetic stimulation (TMS) on the prefrontal cortex and posterior parietal cortex.

DETAILED DESCRIPTION:
The Comprehensive Control Task (CCT) was designed to examine hierarchical control in a single, well-controlled factorial task. On each trial, participants view a letter surrounded by a colored shape at a particular screen location. Color cues the relevant feature, letter or location, for a block of trials. The first trial of a block requires a decision of whether the stimulus is the first position of a circular sequence (sequence start). Subsequent trials require a decision of whether the viewed stimulus follows the previous stimulus in a circular sequence (sequence 1-back). The letter sequence (C-O-M-I-C) and spatial sequence (Top Left-Top Right-Bottom Left-Bottom Right-Top Left) are difficulty-matched.

Shape cues the task to perform. Squares indicate the standard baseline task, and each block begins and ends with baseline trials. Different shapes indicate sub-tasks. In Switching blocks, shape-switches (e.g. from square to circle or circle to square) cue the sequence start task. Shape-repeats cue the sequence 1-back task. In Planning blocks, triangle shapes indicate that the stimulus can be ignored (automatic "no" response). All the while, the last square-shaped stimulus must be retained as a reference for the next square-shaped stimulus. Finally, in Dual blocks, diamond shapes indicate switching (sequence start) and also planning. The reversion back to square shapes requires sequence matching to the distal, previous square.

The design is factorial with stimulus-domain x contextual control x temporal control orthogonally manipulated. Full details of the CCT have been previous described in Nee & D'Esposito, 2016; 2017.

The focus in this study will be comparison of FPl-TMS, MFG-TMS, and S1-TMS in an interleaved fMRI-TMS-fMRI design. The logic is to test the apical status of the FPl/MFG through the extent to which TMS impacts other PFC areas and behavior.

Each experiment will begin with 1 session of the CCT with fMRI to localize PFC targets. Each participant will then perform 3 counter-balanced sessions wherein a different site will be targeted by TMS followed immediately by fMRI on the CCT.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 30
* Right-handed
* Native English speaker or fluent by the age of 6

Exclusion Criteria:

* History of psychiatric disorders
* History of neurological disorders
* Receiving medications for psychiatric or neurological disorders
* Familial history of epilepsy
* Taking any drugs or medications that are pro-epileptic
* Metal anywhere in the head excluding the mouth
* Tinnitus
* Women who are pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek E Nee, PhD, Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Florida State University Psychology Department Building, Tallahassee, Florida
  - FSU MRI Facility, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: Yes
Behavioral and imaging data will be shared
Supporting Information: Analytic Code
Time Frame: Within a year following publication of findings
Access Criteria: Behavioral and imaging data will be accessible from https://nda.nih.gov/edit_collection.html?id=3448 by NDA users.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, participants complete 1) a baseline functional MRI scan to determine targets for transcranial magnetic stimulation, and 2) motor thresholding to determine intensity of transcranial magnetic stimulation. Participants are not assigned to arms if they cannot perform the task inside the MRI scanner (e.g. due to claustrophobia) or if they cannot tolerate transcranial magnetic stimulation.
Groups:
- FPl-TMS Then MFG-TMS Then S1-TMS: Transcranial magnetic stimulation to the lateral frontal pole first followed by middle frontal gyrus followed by primary somatosensory cortex. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- FPl-TMS Then S1-TMS Then MFG-TMS: Transcranial magnetic stimulation to the lateral frontal pole first followed by primary somatosensory cortex followed by middle frontal gyrus. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- MFG-TMS Then FPl-TMS Then S1-TMS: Transcranial magnetic stimulation to the middle frontal gyrus then lateral frontal pole then primary somatosensory cortex. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- MFG-TMS Then S1-TMS Then FPl-TMS: Transcranial magnetic stimulation to the middle frontal gyrus then primary somatosensory cortex then lateral frontal pole. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- S1-TMS Then FPl-TMS Then MFG-TMS: Transcranial magnetic stimulation to primary somatosensory cortex then lateral frontal pole then middle frontal gyrus. Each visit consisted of600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- S1-TMS Then MFG-TMS Then FPl-TMS: Transcranial magnetic stimulation to primary somatosensory cortex then middle frontal gyrus then lateral frontal pole. Each visit consisted of600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
Period: Overall Study
Arm/Group | FPl-TMS Then MFG-TMS Then S1-TMS | FPl-TMS Then S1-TMS Then MFG-TMS | MFG-TMS Then FPl-TMS Then S1-TMS | MFG-TMS Then S1-TMS Then FPl-TMS | S1-TMS Then FPl-TMS Then MFG-TMS | S1-TMS Then MFG-TMS Then FPl-TMS
Started | 6 | 6 | 6 | 9 | 7 | 5
Completed | 6 | 6 | 6 | 6 | 7 | 5
Not Completed | 0 | 0 | 0 | 3 | 0 | 0
Not completed — New piercing could not be removed for scanning | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MFG-TMS Then FPl-TMS Then S1-TMS: Transcranial magnetic stimulation to the middle frontal gyrus first followed by lateral frontal pole followed by primary somatosensory cortex. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- MFG-TMS Then S1-TMS Then FPl-TMS: Transcranial magnetic stimulation to the middle frontal gyrus first followed by primary somatosensory cortex followed by lateral frontal pole. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- S1-TMS Then FPl-TMS Then MFG-TMS: Transcranial magnetic stimulation to primary somatosensory cortex first followed by lateral frontal pole followed by middle frontal gyrus. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- S1-TMS Then MFG-TMS Then FPl-TMS: Transcranial magnetic stimulation to primary somatosensory cortex first followed by middle frontal gyrus followed by lateral frontal pole. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- Total: Total of all reporting groups
Arm/Group | FPl-TMS Then MFG-TMS Then S1-TMS | FPl-TMS Then S1-TMS Then MFG-TMS | MFG-TMS Then FPl-TMS Then S1-TMS | MFG-TMS Then S1-TMS Then FPl-TMS | S1-TMS Then FPl-TMS Then MFG-TMS | S1-TMS Then MFG-TMS Then FPl-TMS | Total
Number analyzed (Participants) | 6 | 6 | 6 | 9 | 7 | 5 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 9 | 7 | 5 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 19 [18 to 21] | 19 [18 to 21] | 19.83 [18 to 25] | 19 [18 to 22] | 19.86 [18 to 21] | 19.8 [18 to 22] | 19.38 [18 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 7 | 3 | 4 | 27
  Male | 3 | 1 | 1 | 2 | 4 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3 | 2 | 2 | 10
  Not Hispanic or Latino | 5 | 5 | 5 | 6 | 5 | 3 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 1 | 3 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 5 | 6 | 8 | 3 | 5 | 31
  More than one race | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 9 | 7 | 5 | 39

OUTCOME MEASURES:

1. Primary Outcome: PFC-PPC Effective Connectivity
Description: effective connectivity among areas of the prefrontal and posterior parietal cortex in the blood oxygenation level dependent (BOLD) signal assessed with functional magnetic resonance imaging (fMRI) [note, this measure has no units, but effective connectivity is a rate measure, so is expressed in Hertz]
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: Participants were included in analysis if they (1) met an 85% overall accuracy on the behavioral task prior to the intervention, (2) completed all three study arms and (3) do not exceed a root mean squared framewise displacement of 0.25, a measure of movement during scans.
Measure: Mean (Standard Error); unit: Hertz
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 30 | 30 | 30
Hertz
  MFG Efferent Connectivity Overall Magnitude | 0.3646 (0.0235) | 0.3756 (0.026) | 0.3425 (0.0237)
  MFG Efferent Connectivity to Temporal Control Areas Magnitude | 0.4519 (0.0367) | 0.466 (0.0404) | 0.4004 (0.0341)
  MFG Efferent Connectivity to Contextual Control Areas Magnitude | 0.2772 (0.0278) | 0.2853 (0.0345) | 0.2846 (0.0295)
  FPl Efferent Connectivity Overall Magnitude | 0.2283 (0.0212) | 0.2352 (0.0232) | 0.2672 (0.0216)
  FPl Efferent Connectivity to Temporal Control Areas Magnitude | 0.3363 (0.0446) | 0.3883 (0.054) | 0.4504 (0.0469)
  FPl Efferent Connectivity to Contextual Areas Magnitude | 0.228 (0.0281) | 0.2184 (0.0287) | 0.2302 (0.0213)
  FPl Efferent Connectivity to Sensorimotor Control Areas Magnitude | 0.1213 (0.0195) | 0.1325 (0.0266) | 0.1948 (0.034)
  MFG Efferent Connectivity Overall Magnitude Change from Baseline | 0.0167 (0.0279) | 0.0277 (0.026) | -0.0054 (0.025)
  MFG Efferent Connectivity to Temporal Control Areas Magnitude Change from Baseline | 0.0442 (0.0393) | 0.0583 (0.0353) | -0.0073 (0.0418)
  MFG Efferent Connectivity to Contextual Control Areas Magnitude Change from Baseline | -0.011 (0.0299) | -0.0029 (0.0341) | -0.0036 (0.0247)
  FPl Efferent Connectivity Overall Magnitude Change from Baseline | 0.0044 (0.0245) | 0.0113 (0.0303) | 0.0433 (0.0272)
  FPl Efferent Connectivity to Temporal Control Areas Magnitude Change from Baseline | 0.035 (0.0512) | 0.087 (0.0613) | 0.1491 (0.0439)
  FPl Efferent Connectivity to Contextual Control Areas Magnitude Change from Baseline | 0.0067 (0.0328) | -0.0029 (0.039) | 0.0089 (0.0377)
  FPl Efferent Connectivity to Sensorimotor Control Areas Magnitude Change from Baseline | -0.033 (0.0262) | -0.0218 (0.0362) | 0.0405 (0.0329)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.5736, ANOVA; The main effect of visit (Baseline, FPl-TMS, MFG-TMS, S1-TMS) on the overall magnitude of MFG efferent connectivity
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.304, ANOVA; Interaction of visit (Baseline, FPl-TMS, MFG-TMS, S1-TMS) and subsystem (Temporal, Contextual Control) on the magnitude of MFG efferent connectivity
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0545, ANOVA; The main effect of visit (Baseline, FPl-TMS, MFG-TMS, S1-TMS) on the overall magnitude of FPl efferent connectivity
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.1134, ANOVA; Interaction of visit (Baseline, FPl-TMS, MFG-TMS, S1-TMS) and Subsystem on the magnitude of FPl efferent connectivity
Statistical Analysis 5: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.4326, ANOVA; The main effect of intervention (FPl-TMS, MFG-TMS, S1-TMS) on the overall magnitude of MFG efferent connectivity
Statistical Analysis 6: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.2546, ANOVA; The interaction of intervention (FPl-TMS, MFG-TMS, S1-TMS) and subsystem (Temporal, Contextual Control) on the magnitude of MFG efferent connectivity
Statistical Analysis 7: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0645, ANOVA; The main effect of intervention (FPl-TMS, MFG-TMS, S1-TMS) on the overall magnitude of FPl efferent connectivity
Statistical Analysis 8: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.2033, ANOVA; Interaction of intervention (FPl-TMS, MFG-TMS, S1-TMS) and Subsystem on the magnitude of FPl efferent connectivity

2. Primary Outcome: PFC-PPC Activation
Description: blood oxygenation level dependent (BOLD) signal in areas of the prefrontal and posterior parietal cortex assessed with functional magnetic resonance imaging (fMRI) [note, this measure has no units]
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: Participants were included in analysis if they (1) met an 85% overall accuracy on the behavioral task prior to the intervention, (2) completed all three study arms and (3) did not exceed a root mean squared framewise displacement of 0.25, a measure of movement during scans.
Measure: Mean (Standard Error); unit: No Unit
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 31 | 31 | 31
No Unit
  Overall BOLD | 0.1132 (0.0313) | 0.1155 (0.0227) | 0.0992 (0.0274)
  Overall BOLD in Temporal Control BOLD Subsystem | 0.1519 (0.0425) | 0.1619 (0.031) | 0.162 (0.0357)
  Overall BOLD in Contextual Control Subsystem | 0.1499 (0.0393) | 0.1667 (0.0289) | 0.1253 (0.034)
  Overall BOLD in Sensorimotor Control Subsystem | 0.15 (0.0396) | 0.1143 (0.0322) | 0.0998 (0.0291)
  Temporal Control BOLD in Temporal Control Subsystem | 0.2269 (0.0361) | 0.305 (0.0337) | 0.2531 (0.0379)
  Temporal Control BOLD in Contextual Control Subsystem | 0.038 (0.0327) | 0.1167 (0.0319) | 0.0802 (0.0328)
  Temporal Control BOLD in Sensorimotor Control Subsystem | -0.0086 (0.0323) | 0.0621 (0.0334) | -0.0186 (0.031)
  Contextual Control BOLD in Temporal Control Subsystem | 0.1719 (0.0382) | 0.1542 (0.0387) | 0.1535 (0.0329)
  Contextual Control BOLD in Contextual Control Subsystem | 0.3773 (0.0342) | 0.331 (0.037) | 0.349 (0.0352)
  Contextual Control BOLD in Sensorimotor Control Subsystem | 0.3079 (0.0256) | 0.3133 (0.0315) | 0.3008 (0.0298)
  Temporal x Contextual Control BOLD in Temporal Control Subsystem | -0.0717 (0.0366) | -0.065 (0.0346) | -0.0177 (0.0461)
  Temporal x Contextual Control BOLD in Contextual Control Subsystem | 0.2218 (0.0333) | 0.1645 (0.0357) | 0.2455 (0.0365)
  Temporal x Contextual Control BOLD in Sensorimotor Control Subsystem | 0.2713 (0.0379) | 0.2402 (0.0376) | 0.2666 (0.0283)
  Overall BOLD Change from Baseline | 0.0096 (0.0267) | 0.0120 (0.0239) | -0.0044 (0.0272)
  Overall BOLD in Temporal Control Subsystem Change from Baseline | -0.0336 (0.0344) | -0.0236 (0.0317) | -0.0235 (0.0333)
  Overall BOLD in Contextual Control Subsystem Change from Baseline | 0.0187 (0.0333) | 0.0355 (0.0289) | -0.0059 (0.0308)
  Overall BOLD in Sensorimotor Control Subsystem Change from Baseline | 0.0777 (0.0348) | 0.042 (0.0302) | 0.0275 (0.0314)
  Temporal Control BOLD in Temporal Control Subsystem Change from Baseline | -0.0783 (0.0352) | -0.0002 (0.0343) | -0.0521 (0.0391)
  Temporal Control BOLD in Contextual Control Subsystem Change from Baseline | 0.0067 (0.027) | 0.0854 (0.0311) | 0.0489 (0.0398)
  Temporal Control BOLD in Sensorimotor Control Subsystem Change from Baseline | 0.06 (0.0303) | 0.1307 (0.0321) | 0.05 (0.0388)
  Contextual Control BOLD in Temporal Control Subsystem Change from Baseline | 0.028 (0.0405) | 0.0103 (0.0417) | 0.0096 (0.0398)
  Contextual Control BOLD in Contextual Control Subsystem Change from Baseline | -0.0228 (0.0347) | -0.0691 (0.0262) | -0.0511 (0.0274)
  Contextual Control BOLD in Sensorimotor Control Subsystem Change from Baseline | -0.0498 (0.033) | -0.0444 (0.0257) | -0.0569 (0.0265)
  Temporal x Contextual Control BOLD in Temporal Control Subsystem Change from Baseline | 0.0194 (0.0386) | 0.0261 (0.0369) | 0.0734 (0.041)
  Temporal x Contextual Control BOLD in Contextual Control Subsystem Change from Baseline | 0.0797 (0.0364) | 0.0224 (0.0388) | 0.1034 (0.0315)
  Temporal x Contextual Control BOLD in Sensorimotor Control Subsystem Change from Baseline | 0.0564 (0.0348) | 0.0253 (0.0446) | 0.0517 (0.0306)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.8152, ANOVA; Main effect of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) on overall BOLD actviation
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0085, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) and subsystem (temporal, contextual, sensorimotor control) on overall BOLD activation
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.1551, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) and temporal control on BOLD activation
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.6431, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) and contextual control on BOLD activation
Statistical Analysis 5: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.2447, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), temporal control, and contextual control on BOLD activation
Statistical Analysis 6: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0002, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), temporal control, and subsystem (temporal, contextual, sensorimotor) on BOLD activation
Statistical Analysis 7: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.1339, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), contextual control, and subsystem on BOLD activation
Statistical Analysis 8: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.1315, ANOVA; Interaction of visit, temporal control, contextual control, and subsystem on BOLD activation
Statistical Analysis 9: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.6836, ANOVA; The main effect of intervention arm (FPl-TMS, MFG-TMS, S1-TMS) on overall BOLD activation
Statistical Analysis 10: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.2146, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1-cTBS) and subsystem (temporal, contextual, sensorimotor control) on overall BOLD activation
Statistical Analysis 11: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.1541, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1-cTBS) and temporal control on BOLD activation
Statistical Analysis 12: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.6657, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1-cTBS) and contextual control on BOLD activation
Statistical Analysis 13: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.5619, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), temporal control, and contextual control on BOLD activation
Statistical Analysis 14: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.5148, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), temporal control, and subsystem (temporal, contextual, sensorimotor) on BOLD activation
Statistical Analysis 15: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.5428, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), contextual control, and subsystem (temporal, contextual, sensorimotor) on BOLD activation
Statistical Analysis 16: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.1249, ANOVA; Interaction of intervention, temporal control, contextual control, and subsystem on BOLD activation

3. Secondary Outcome: Temporal Control Performance (Error Rate)
Description: behavioral performance (error rate) on conditions involving temporal control in the comprehensive control task
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: Participants were included in analysis if they (1) met an 85% overall accuracy on the behavioral task prior to the intervention, and (2) completed all three study arms.
Measure: Mean (Standard Error); unit: Error Rate (%)
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 32 | 32 | 32
Error Rate (%)
  Difference between high and low temporal control trials error rate | 4.541 (1.043) | 3.826 (0.999) | 4.329 (1.121)
  Difference between high and low temporal control subtask trial error rate | -0.293 (0.490) | -0.942 (0.683) | 0.358 (0.340)
  Difference between high and low temporal control return trial error rate | 9.375 (2.108) | 8.594 (2.011) | 8.301 (2.221)
  Difference between high and low temporal control trials error rate relative to baseline | 0.042 (1.454) | -0.673 (1.450) | -0.169 (1.415)
  Difference between high and low temporal control subtask trial error rate relative to baseline | 0.769 (0.697) | 0.119 (0.898) | 1.420 (0.512)
  Difference between high and low temporal control return trial accuracy relative to error rate | -0.684 (3.075) | -1.465 (2.620) | -1.758 (2.717)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.9504, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) and temporal control on error rate
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.7318, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), and temporal control on error rate
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.8424, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS) and temporal control on error rate
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.7652, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), and temporal control on error rate

4. Secondary Outcome: Contextual Control Performance (Error Rate)
Description: behavioral performance (error rate) on conditions involving contextual control in the comprehensive control task
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Error rate (%)
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 32 | 32 | 32
Error rate (%)
  Difference between high and low contextual control trials error rate | 5.580 (1.240) | 6.950 (1.200) | 5.890 (1.210)
  Difference between high and low contextual control subtask trial error rate | 1.990 (0.360) | 2.960 (0.580) | 2.700 (0.510)
  Difference between high and low contextual control return trial error rate | 9.180 (2.412) | 10.940 (2.240) | 9.080 (2.378)
  Difference between high and low contextual control error rate relative to baseline | 2.030 (0.922) | 3.400 (1.100) | 2.340 (1.365)
  Difference between high and low contextual control subtask trial error rate relative to baseline | 0.270 (0.410) | 1.240 (0.577) | 0.980 (0.596)
  Difference between high and low contextual control return trial error rate relative to baseline | 3.810 (1.846) | 5.570 (2.089) | 3.710 (2.690)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0266, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) and contextual control on error rate
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.2386, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return) and contextual control on error rate
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.4211, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS) and contextual control on error rate
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.7503, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return) and contextual control on error rate

5. Secondary Outcome: Temporal x Contextual Control Performance (Error Rate)
Description: behavioral performance (error rate) of the interaction of temporal and contextual control in the comprehensive control task
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Error rate (%)
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 32 | 32 | 32
Error rate (%)
  Interaction contrast of temporal and contextual control on error rate | -1.810 (1.098) | 0.082 (1.151) | -2.181 (1.095)
  Interaction contrast of temporal and contextual control on error rate in sub-task trials | 1.270 (0.453) | 1.141 (0.594) | 1.400 (0.400)
  Interaction contrast of temporal and contextual control on error rate in return trials | -4.880 (2.319) | -0.977 (2.199) | -5.762 (2.127)
  Interaction contrast of temporal and contextual control on error rate relative to baseline | 2.210 (1.052) | 4.102 (1.430) | 1.839 (1.093)
  Interaction contrast of temporal and contextual control on error rate in sub-task trials vs baseline | 0.030 (0.649) | -0.099 (0.708) | 0.160 (0.488)
  Interaction contrast of temporal and contextual control on error rate in return trials vs baseline | 4.400 (2.043) | 8.303 (2.608) | 3.518 (2.057)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0091, ANOVA; Interaction of Visit (Baseline, MFG-cTBS, FPl-cTBS, S1), Temporal Control, and Contextual Control on error rate
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0045, ANOVA; Interaction of Visit (Baseline, MFG-cTBS, FPl-cTBS, S1), phase (sub-task, return), Temporal Control, and Contextual Control on error rate
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.1082, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1), Temporal Control, and Contextual Control on error rate
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0659, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1), phase (sub-task, return), Temporal Control, and Contextual Control on error rate

6. Secondary Outcome: Temporal Control Performance (Reaction Time)
Description: behavioral performance (reaction time in milliseconds) on conditions involving temporal control in the comprehensive control task
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 32 | 32 | 32
Milliseconds
  Difference between high and low temporal control trial reaction time | 15.700 (10.162) | 11.987 (10.200) | -2.244 (10.872)
  Difference between high and low temporal control subtask trial reaction time | -18.172 (7.985) | -16.540 (7.435) | -23.348 (9.823)
  Difference between high and low temporal control return trial reaction time | 49.577 (18.654) | 40.514 (16.972) | 18.861 (17.568)
  Difference between high and low temporal control trial reaction time relative to baseline | 37.631 (12.288) | 33.917 (14.750) | 19.687 (13.650)
  Difference between high and low temporal control subtask trial reaction time relative to baseline | 43.256 (9.600) | 44.888 (13.390) | 38.080 (14.470)
  Difference between high and low temporal control return trial reaction time relative to baseline | 32.010 (20.900) | 22.947 (26.980) | 1.294 (21.600)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0211, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) and temporal control in reaction time
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.4964, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), and temporal control in reaction time
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.3129, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS) and temporal control in reaction time
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.5439, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), and temporal control in reaction time

7. Secondary Outcome: Contextual Control Performance (Reaction Time)
Description: behavioral performance (reaction time in milliseconds) on conditions involving contextual control in the comprehensive control task
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 32 | 32 | 32
Milliseconds
  Difference between high and low contextual control trial reaction time | 197.700 (16.600) | 185.443 (14.300) | 160.900 (10.600)
  Difference between high and low contextual control subtask trial reaction time | 163.774 (16.500) | 146.982 (13.300) | 132.500 (9.877)
  Difference between high and low contextual control return trial reaction time | 231.652 (20.400) | 223.900 (19.300) | 189.270 (18.278)
  Difference between high and low contextual control trial reaction time relative to baseline | -0.700 (17.500) | -12.957 (12.200) | -37.500 (13.400)
  Difference between high and low contextual control subtask trial reaction time relative to baseline | -13.982 (14.660) | -30.773 (11.757) | -45.256 (12.360)
  Difference between high and low contextual control return trial reaction time relative to baseline | 12.610 (26.500) | 4.858 (21.700) | -29.772 (23.500)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0344, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS) and contextual control in reaction time
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.5113, ANOVA; Interaction between visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), and contextual control in reaction time
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0301, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS) and contextual control in reaction time
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.6931, ANOVA; Interaction between intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), and contextual control in reaction time

8. Secondary Outcome: Temporal Control x Contextual Control Performance (Reaction Time)
Description: behavioral performance (reaction time in milliseconds) on the interaction between temporal control and contextual control in the comprehensive control task
Time Frame: baseline, pre-intervention and immediately after intervention (5 minutes to 1 hour post-TMS)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
Number analyzed (Participants) | 32 | 32 | 32
Milliseconds
  Interaction contrast of temporal control x contextual control trials on reaction time | 55.600 (8.500) | 53.162 (10.800) | 53.280 (9.200)
  Interaction contrast of temporal control x contextual control subtask trials on reaction time | 141.900 (12.700) | 131.227 (16.300) | 125.100 (10.100)
  Interaction contrast of temporal control x contextual control return trials on reaction time | -30.697 (12.100) | -24.903 (15.700) | -18.547 (14.800)
  Interaction contrast of temporal control x contextual control trials on reaction time vs baseline | 32.200 (11.800) | 29.762 (13.160) | 29.880 (10.399)
  Interaction contrast of temporal control x contextual control subtask trials on RT vs baseline | 14.614 (12.160) | 3.941 (15.180) | -2.186 (12.800)
  Interaction contrast of temporal control x contextual control return trials on RT vs baseline | 49.703 (22.550) | 55.497 (24.400) | 61.853 (21.600)
Statistical Analysis 1: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0189, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), temporal control, and contextual control on reaction time
Statistical Analysis 2: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.0763, ANOVA; Interaction of visit (Baseline, MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), temporal control, and contextual control on reaction time
Statistical Analysis 3: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.9701, ANOVA; Interaction of intervention (MFG-cTBS, FPl-cTBS, S1-cTBS), temporal control, and contextual control on reaction time
Statistical Analysis 4: Comparison: FPl-TMS vs MFG-TMS vs S1-TMS; Test type: Superiority; p = 0.3826, ANOVA; Interaction of intervention(MFG-cTBS, FPl-cTBS, S1-cTBS), phase (sub-task, return), temporal control, and contextual control on reaction time

ADVERSE EVENTS:
Time Frame: 1 month (this is the duration over which each participant was monitored for adverse events)
Groups:
- FPl-TMS: Transcranial magnetic stimulation to the lateral frontal pole. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- MFG-TMS: Transcranial magnetic stimulation to the middle frontal gyrus. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
- S1-TMS: Transcranial magnetic stimulation to primary somatosensory cortex. Each visit consists of 600 pulses delivered in 50 Hz bursts every 5 Hz for 40 seconds at 80% of active motor threshold to one target.
  transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance.
Arm/Group | FPl-TMS | MFG-TMS | S1-TMS
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 1/37 | 0/37 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FPl-TMS (N=37) | MFG-TMS (N=37) | S1-TMS (N=38)
Mild vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Subject experienced mild vertigo following TMS. The issue resolved within five minutes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT04464473/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04464473/ICF_001.pdf